CLINICAL TRIAL: NCT02677428
Title: Remotely-Delivered Benefits Counseling for Service Connection Applicants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1319-R
Record Dates: First submitted 2016-01-22; First posted 2016-02-09 (Estimated); Results first posted 2020-08-03 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Job Satisfaction; Unemployment
Keywords: Veterans; world wide web; Counseling; Workman's Compensation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remotely Delivered Benefits Counseling (Experimental): Veterans will complete three intervention modules online. For the first module, Veterans will be instructed on how to use the website and its purpose; will be asked about their perception of the relationship between disability benefits and work. An explanation of relationship between disability benefits and work will be provided. For the second module, Veterans' feelings and attitudes towards employment will be solicited. Motivational Interviewing exercises will be implemented; barriers to work including the disabling condition and consideration of treatment for disabling conditions will be reviewed. An action plan will be developed. For the third module, inquiries will be made regarding the Veteran's reaction to the service-connection decision; information will be provided on how to appeal the decision. Veterans will be asked to reconsider work and financial goals in light of service-connection award. Their action plan will be reviewed. Follow-up resources will be provided.
  Interventions: Behavioral: Remotely-Delivered Benefits Counseling
- Control (Active Comparator): The control condition will involve referrals to VA websites and represents enhanced treatment-as-usual. A Veteran who completes a Compensation examination ordinarily has no further treatment or referral as part of the Compensation examination. The information about benefits-related websites controls for having information available about benefits and receiving encouragement to pursue that information. The control condition involves being urged to explore links to three VA websites with Compensation & Pension-related information: (a) the Veterans Benefits Administration (VBA) website with links about VA disability compensation, (b) the VBA site with fact sheets about the different types of benefits available to Veterans, and (c) the VBA websites for the local C&P office where issues pertaining to an individual Veteran's specific application are addressed.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Remotely-Delivered Benefits Counseling — Veterans will complete three intervention modules online. For the first module, Veterans will be instructed on how to use the website and its purpose; will be asked about their perception of the relationship between disability benefits and work. An explanation of relationship between disability benefits and work will be provided. For the second module, Veterans' feelings and attitudes towards employment will be solicited. Motivational Interviewing exercises will be implemented; barriers to work including the disabling condition and consideration of treatment for disabling conditions will be reviewed. An action plan will be developed. For the third module, inquiries will be made regarding the Veteran's reaction to the service-connection decision; information will be provided on how to appeal the decision. Veterans will be asked to reconsider work and financial goals in light of service-connection award. Their action plan will be reviewed. Follow-up resources will be provided.
  Arms: Remotely Delivered Benefits Counseling
Behavioral: Control — The control condition will involve referrals to VA websites and represents enhanced treatment-as-usual. A Veteran who completes a Compensation examination ordinarily has no further treatment or referral as part of the Compensation examination. The information about benefits-related websites controls for having information available about benefits and receiving encouragement to pursue that information. The control condition involves being urged to explore links to three VA websites with Compensation & Pension-related information: (a) the VBA website with links about VA disability compensation, (b) the VBA site with fact sheets about the different types of benefits available to Veterans, and (c) the VBA websites for the local C&P office where issues pertaining to an individual Veteran's specific application are addressed.
  Arms: Control

SUMMARY:
A significant portion of Veterans who apply for disability benefits have difficulty finding and sustaining employment, and are concerned that working for pay will jeopardize their receipt of service-connection benefits. In a completed clinical trial, Veterans who received Motivational Interview-formatted counseled about opportunities to work and receive service-connection went on to work for pay significantly more often than controls. The proposed clinical trial will test this counseling's efficacy when it is delivered by an automated computer program.

DETAILED DESCRIPTION:
Current application rates suggest that more than half of Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Veterans will eventually apply for some form of service-connection, with approximately 100,000 Veterans per year being evaluated for psychiatric conditions. Veterans applying for service-connection for psychiatric conditions are in distress, and often are having occupational difficulties, but these are unaddressed during a typical Compensation and Pension evaluation. Counseling that addresses beneficiaries' concerns about losing compensation payments if working for pay, when supplemented by vocational supports, has been associated with increased employment among people disabled by chronic psychiatric conditions. This group has developed an online Benefits Counseling intervention tailored to help Veterans applying for service-connection engage in work-related activities. The investigators have demonstrated the efficacy of a face-to-face version of Benefits Counseling in a completed Rehabilitation Research & Development-funded six-month clinical trial in which Veterans assigned to Benefits Counseling worked significantly more days than controls,(p<.05, effect size = 0.69), reflecting an average of three more days of employment at six month follow-up. The investigators then used a supplement from Rehabilitation Research & Development to develop a web-based version of this counseling, so that the counseling could be delivered without a counselor on-site. The web-based intervention was modified based on user feedback, but the extent to which it will be used by Veterans at home and how it will impact their behavior is unknown. In the proposed clinical trial, Veterans working two or fewer days per week who are presenting for a Compensation & Pension examination for a psychiatric disorder will be assessed at baseline and then urged to log in afterwards to a website for random assignment to either Remotely-Delivered Benefits Counseling (n=65) or Veterans Benefits Administration web sites (n=65), and will then be assessed at 4, 12, and 24 weeks after randomization in order to calculate standardized group mean differences between the slopes over time. The primary outcome measure will be the treatment-by-time slope of hours of paid work. Exploratory analyses will estimate associations of potential mediators of treatment response with this outcome. The proposed study will provide estimates of the efficacy of remotely-delivered Benefits Counseling initiated at Compensation and Pension examinations, a widely-used point of contact with VA.

ELIGIBILITY:
Inclusion Criteria:

* All enrolled participants will have difficulty working as evidenced by a "Yes" response to any sub-part of the following question:

  * During the past 4 weeks, have you had any of the following problems with your work or other regular daily activities as a result of any emotional problems (such as feeling depressed or anxious):

    * (a) Cut down on the amount of time you spent on work or other activities?
    * (b) Accomplished less than you would like?
    * (c) Didn't do work or other activities as carefully as usual?
* Participants will also meet the following inclusion criteria:

  * i. A Compensation and Pension evaluation by a psychiatrist or psychologist is scheduled
  * ii. Does not have a service-connected physical disability rated over 30%
  * iii. Is not service-connected for a psychiatric condition (0% service-connection is allowed, as Veterans with 0% service-connection have not received any benefit payments)
  * iv. Age 18-65
  * v. Reports access to an internet-connected computer/tablet and a working telephone
  * vi. Reports working an average of two or fewer days per week for pay over the preceding 4 weeks
  * vii. Self-reported ability to participate psychologically and physically, able to give informed consent and complete assessments; viii. Reports being able to read (this is necessary for understanding the website)
  * ix. Expressed interest in sampling whatever website is provided

Exclusion Criteria:

* Already receiving Supplemental Security Income (SSI) or Social Security Disability Insurance (SSDI)
* Has a conservator

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc I. Rosen, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Central Western Massachusetts Healthcare System, Leeds, MA, Leeds, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Only with a data sharing agreement. There is no provision for data sharing in the approved IRB protocol.
Supporting Information: Study Protocol, ICF
Time Frame: By June 2020.
Access Criteria: After a data sharing agreement has been entered into. The plan will specify the requester, purpose, and agreement to keep the data confidential and not disclose it further.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two VA Medical Centers in New England between December 2015 and December 2018. 32 participants who consented to the study did not log into the study website and were thus excluded from analysis.
Groups:
- Control Website: The control website will involve a webpage containing referrals to VA websites and represents enhanced treatment-as-usual. A Veteran who completes a Compensation examination ordinarily has no further treatment or referral as part of the Compensation examination. The information provided on the control website controls for having information available about benefits and receiving encouragement to pursue that information. The control condition involves being urged to explore links to three VA websites with Compensation & Pension-related information: (a) the Veterans Benefits Administration (VBA) website with links about VA disability compensation, (b) the VBA site with fact sheets about the different types of benefits available to Veterans, and (c) the VBA websites for the local C&P office where issues pertaining to an individual Veteran's specific application are addressed.
Period: Overall Study
Arm/Group | Remotely Delivered Benefits Counseling | Control Website
Started | 63 | 55
Completed | 63 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: The control website will involve a webpage containing referrals to VA websites and represents enhanced treatment-as-usual. A Veteran who completes a Compensation examination ordinarily has no further treatment or referral as part of the Compensation examination. The information provided on the control website controls for having information available about benefits and receiving encouragement to pursue that information. The control condition involves being urged to explore links to three VA websites with Compensation & Pension-related information: (a) the Veterans Benefits Administration (VBA) website with links about VA disability compensation, (b) the VBA site with fact sheets about the different types of benefits available to Veterans, and (c) the VBA websites for the local C&P office where issues pertaining to an individual Veteran's specific application are addressed.
- Total: Total of all reporting groups
Arm/Group | Remotely Delivered Benefits Counseling | Control | Total
Number analyzed (Participants) | 63 | 55 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (12.6) | 41.1 (11.0) | 39.8 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 49 | 44 | 93
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 41 | 36 | 77
  Race/Ethnicity: Hispanic | 12 | 10 | 22
  Race/Ethnicity: Black | 5 | 7 | 12
  Race/Ethnicity: Other | 5 | 2 | 7
Problematic Substance Use [Count of Participants; unit: Participants] | 41 | 37 | 78
Provisional PTSD Diagnosis [Count of Participants; unit: Participants] | 41 | 38 | 79
Brief Severity Index [Mean (Standard Deviation); unit: units on a scale] — The BSI is a self-reported measure of psychological distress. It is composed of 53 items from nine primary symptom dimensions. Each item is rated on a 5 point Likert scale of distress (0 "not at all" to 4 "extremely").
  The global severity index is calculated by summing all items and then dividing by the total number of items endorsed, so higher scores indicate more distress.
  The Depression dimension is calculated by summing the six items in this dimension and then dividing by number of items endorsed, so higher scores indicate more distress on this dimension.
  units on a scale
    Global Severity index | 1.6 (.7) | 1.4 (.6) | 1.5 (.7)
    Depression subscale | 1.6 (1.0) | 1.7 (.9) | 1.7 (.9)
Competitive Work [Mean (Standard Deviation); unit: hours per week] — Competitive work is work done for pay that is not sponsored by a treatment or other program. Examples include cashier, day laborer, cook at a restaurant, military service.
  hours per week | 2.8 (6.6) | 2.0 (5.1) | 2.4 (6.0)
Any work-related activities [Mean (Standard Deviation); unit: days per month] — Work-related activities is a sum of days engaged in any of the following work categories: supervised work (work with onsite training or close supervision eg. peer mentoring program, easter seals work program); competitive work (work for pay); vocational rehabilitation (unpaid vocational rehabilitation eg. Marrakech, WAGE, Social Skills Training); School (community college, GED coursework, vocational training, technical training); Volunteer work; Illicit work (eg. panhandling, selling drugs); Other types of work.
  days per month | 7.4 (8.1) | 5.8 (7.4) | 6.7 (7.8)
Income, past 28 days [Mean (Standard Deviation); unit: dollars] | 1790 (1730) | 2318 (2498) | 2036 (2130)

OUTCOME MEASURES:

1. Primary Outcome: Hours Per Week of Paid Work
Description: This calendar measure will be used to determine whether, and on what days the Veteran engaged in paid work activities.
Time Frame: Assessed at baseline, and 4, 12 and 24 weeks post-randomization. Each assessment is for the period since prior assessment
Measure: Mean (Standard Deviation); unit: hours per week
Arm/Group | Remotely Delivered Benefits Counseling | Control
Number analyzed (Participants) | 63 | 55
hours per week
  Baseline | 2.8 (6.6) | 2.0 (5.1)
  Week 4 | 4.8 (10.7) | 4.0 (10.7)
  Week 12 | 6.8 (14.6) | 5.6 (12.8)
  Week 24 | 9.6 (19.5) | 7.0 (14.1)

2. Secondary Outcome: Work Importance and Confidence Ruler
Description: This measure consists of six questions about respondent's ability to work to his/her "fullest capacity" currently, how ready they are to work to fullest capacity, how important it is to work to fullest capacity, how important it is to work for pay, and how confident one in in ability work to fullest capacity. Items are rated on an 11 point Likert scale, ranging from 0 to 10, with higher scores indicating more importance (0 "not at all important" to 10 "very important") and more confidence (0 "not at all confident" to 10 "completely confident") in one's ability. We report the mean/median of the scores (range 0-10) at each timepoint by treatment group.
  This measure has been used to show that Veteran-rated importance of work was associated with engagement in Compensated Work Therapy among Veterans with vocational and psychiatric difficulties. It was collected at Baseline, Week 4, Week 12 and week 24.
Time Frame: as for outcome 1
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Remotely Delivered Benefits Counseling | Control
Number analyzed (Participants) | 63 | 55
units on a scale
  Baseline | 7.03 (1.81) | 6.72 (2.57)
  Week 4 | 7.17 (2.02) | 7.08 (1.98)
  Week 12 | 7.34 (1.99) | 7.28 (2.32)
  Week 24 | 7.42 (1.76) | 7.54 (2.19)

ADVERSE EVENTS:
Time Frame: 24 weeks (study participation)
Arm/Group | Remotely Delivered Benefits Counseling | Control
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/63 | 1/55
Other Adverse Events (participants affected / at risk) | 0/63 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remotely Delivered Benefits Counseling (N=63) | Control (N=55)
Suicide Risk (Psychiatric disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT02677428/Prot_SAP_000.pdf
  • Informed Consent Form (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT02677428/ICF_001.pdf